CLINICAL TRIAL: NCT00952471
Title: Reduction in Clinical Variance Using Targeted Design Changes in Computerized Provider Order Entry Order (CPOE) Sets
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brian Jacobs (Other)
Collaborators: Siemens Medical (Unknown)
Responsible Party: Sponsor-Investigator, Brian Jacobs, MD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 05-11-34
Record Dates: First submitted 2009-07-24; First posted 2009-08-06 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Asthma Exacerbation
Keywords: Asthma; Children; CPOE; Decision Support; Framing; Heuristic; Order Sets
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baseline Period (No Intervention): Patients in the baseline period were cared for using the standard historical electronic order set.
- Post Intervention Period (Active Comparator): Patients in the Post intervention period were cared for with evidence-bsed modified order set changes
  Interventions: Other: Evidence Based Intervention to order set

INTERVENTIONS:
Other: Evidence Based Intervention to order set — The order set was altered to include evidence based care items
  Arms: Post Intervention Period

SUMMARY:
Selective redesign of order sets using different ways to frame the order and physician decision-making in a computerized provider order entry system could increase adherence to evidence-based care and reduce population-specific variance.

DETAILED DESCRIPTION:
Variance in ordering of care can be characterized as the lack of uniform use of specific treatments by clinicians for a given medical condition. Unwarranted variance in healthcare has been associated with prolonged length of stay, diminished health and increased cost. Practice variation in the management of asthma can be significant and few investigators have evaluated strategies to reduce this variation. We hypothesized that selective redesign of order sets using different ways to frame the order and physician decision-making in a computerized provider order entry system could increase adherence to evidence-based care and reduce population-specific variance.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted using an acute asthma exacerbation order set.

Exclusion Criteria:

* Patients who did not have either an admission or discharge diagnosis of asthma exacerbation.
* In addition, patients admitted to the intensive care unit directly or transferred to the intensive care unit within 24-hours were excluded from analysis.
* Finally, patients were excluded from analysis if asthma was not the presenting problem.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2004-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Reduced variation from in evidence-based care through integrating evidence into the clinician workflow in the EMR system. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States